CLINICAL TRIAL: NCT04519203
Title: The Use of Surgical Pleth Index in Guiding Anesthesia in Gastroenterological Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: general electric healthcare Finland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R20006
Record Dates: First submitted 2020-02-21; First posted 2020-08-19 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2021-04

CONDITIONS: Intraoperative Complications; Intraoperative Hypotension; Intraoperative Hypertension
Keywords: Nociception; Intraoperative monitoring; Surgical pleth index
MeSH Terms: conditions — Intraoperative Complications | interventions — Reference Standards

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients are randomized using sealed envelopes. The ramdomization will be kept blinded to the study subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SPI group (Active Comparator): Group of patients where opioid consumption will be guided using SPI target
  Interventions: Device: SPI
- Control Group (Active Comparator): Group of patients where only standard monitoring and patient reaction will be used to guide opioid administration during intraoperative period
  Interventions: Device: Standard

INTERVENTIONS:
Device: SPI — Either standard monitoring alone or added with SPI
  Arms: SPI group
Device: Standard — Standard monitoring alone
  Arms: Control Group

SUMMARY:
Surgical Pleth Index (SPI) is an intraoperative monitor aimed into detection of nociception and guidance of intraoperative opioid administration. Using such a device opioid administration could be potentially optimized during intraoperative period. this study will aim to show whether SPI could be used to reduce unwanted events and lower opioid consumption in gastroenterological surgery. The study will be blinded and randomized including two study arms with either SPI monitoring included or standard monitoring alone.

DETAILED DESCRIPTION:
Patients are extensively monitored intraoperatively. Even though there are monitors for the measurement of nociception, it has not gained wide acceptance partly because of limited and scarce evidence on the efficacy and optimal use. Especially elderly patients undergoing major operation might benefit from optimization of opioid administration. Surgical Pleth Index (SPI) is an intraoperative monitoring aimed for detection of nociceptive stimulus.

The aim of this research is to study whether SPI could be used to guide opioid administration in gastroenterological surgery. The study will consist of a total 80 patients which are randomized into two groups. The study sample is based on power calculation for the reduction of remifentanil consumption.

In the study group the opioid administration will be guided using a SPI based protocol. In the control group the opioid administration will be based on standard monitoring and clinical decision alone. The aim of the study will be to study whether opioid administration optimized using SPI can lover need for anticholinergic drugs, reduce need for opioids or diminish the amount of unwanted side effects postoperatively. The patients will be treated using target controlled infusions of remifentanil and propofol.

The data will be collected intraoperatively using electronic software and using a study data collection form by study personel. All study procedures will take place during operative period.

The study power was calculated using a study comparing depth of anesthesia and depth of nociception balance-controlled group into a group without these monitors. In the group with monitoring the consumption of remifentanil was 9,5±3.8 mg/kg/h while in the unmonitored group the consumption was 12.3 mg/kg/h(Chen, 2010). While taking into notice α= 0,005 and β=90% a number of 39 patients in each group is needed. Based on these we chose 80 patients to be included in the study.

All collected data will be used into statistical analysis ass applicable. Statistical analysis plan describing the analytical principles and statistical techniques to be employed in order to address the primary and secondary objectives, as specified in the study protocol or plan.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide a written informed consent
* Age 50 years or above
* Laparoscopic or laparotomic surgery requiring intubation with an expected intraoperative time at least two hours.
* ASA classification 1-3

Exclusion Criteria:

* Implanted cardiac pacemaker or known condition with irregular heart rate at the time of inclusion or induction
* Chronic use of opioids
* BMI >35
* Known allergy for study medications
* Over 5 extrasystoles per minute at the time of induction or inclusion
* The use of epidural catheter during the last one hour before surgery or need for catheter intraoperatively (if new catheter is placed at the beginning of surgery test dosage may be used without the need for patient exclusion)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Intraoperative remifentanil consumption | intraoperative time
  The consumption of the remifentanil intraoperatively

SECONDARY OUTCOMES:
severe hypotension | intraoperative time
  MAP <55 mmHg, or -30% from the baseline value
intermediate hypotension | intraoperative time
  MAP <65 mmHg, or -20% from the baseline value
hypertension | intraoperative time
  RRsys >140 mmHg or +20 % from baseline value
Bradycardia | intraoperative time
  Heart rate<45
tachycardia | intraoperative time
  Heart rate>90
Inraoperative propofol consumption | intraoperative time
Desorientation/ grade of sedation during postoperative care treatment | 2-4 hours
  The postoperative desoroentation during immediate post-operative period at postanesthesia care unit. Measured using modified aldrete score
Postoperative nausea and vomiting | 2-4 hours
  The postoperative nausea and vomiting during immediate post-operative period at postanesthesia care unit. Measured using modified aldrete score.
Postoperative opioid consumption | 2-4 hours
  The postoperative opioid consumption during immediate post-operative period at postanesthesia care unit.
Fading of intraoperative relaxation | intraoperative time
  The characteristics of intraoperative relaxation using EMG measurement

CONTACTS AND LOCATIONS:
Overall Officials: Jarkko Harju, MD, PhD, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No